CLINICAL TRIAL: NCT05388344
Title: LUMINA : Measure the Effectiveness of the Booklet Named "Comprendre Les Essais Cliniques" With Patients Included or Not Included in Clinical Trials Within the Clinical Neurosciences - Rheumatology Pole of the CHU de Nice
Brief Title: LUMINA : Measure the Effectiveness of the Booklet Named "Comprendre Les Essais Cliniques"
Acronym: LUMINA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Neuro03
Record Dates: First submitted 2021-09-24; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Rheumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Booklet reading — Submission of the questionnaire before and after booklet reading

SUMMARY:
Various studies have shown that many patients do not understand all the information provided by the study investigator and by the information sheet before entering a clinical research protocol. Many materials has been developped in previous research, trying to improve patients' understanding. Nonetheless, their effectiveness remains uncertain.

The "LUMINA" project aims to measure the effectiveness of the booklet named "Comprendre les essais cliniques" with patients included or not included in clinical trials within the Clinical Neurosciences - Rheumatology pole of the CHU de Nice. The design of this study is "before/after". A questionnaire was submitted to the patients before and after reading the booklet. That method is used in order to show if there was a difference between the score obtained from the questionnaire before and after reading. This difference could reflect an improvement in patients' comprehension and, by extension, the effectiveness of the support the team developed.

ELIGIBILITY:
Inclusion Criteria:

* age <18
* patient coming for a consultation or an hospitalization within the Clinical Neurosciences-Rheumatology pole of the CHU de Nice, or companions/caregivers who helps the patients understand
* Patient able to read and to understand the french language,
* Patient included or not in clinical trials.

Exclusion Criteria:

* Participants unable to read
* Patient unable to understand the french language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants coming for a consultation or an hospitalization within the Clinical Neurosciences-Rheumatology pole of the CHU de Nice
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the booklet | day 1
  Measurement of the score (0 to 13)obtained from the assessment questionnaire (right or wrong) created for the study, before and after reading the booklet right = 1 point, wrong = 0 point . Score: points addition

SECONDARY OUTCOMES:
Assess the booklet's lisibility | day 1
  Calculate the "Flesch Reading ease" index of the booklet
Assess the difference in understanding between patient groups | day 1
  Measurement of the impact of different variables, such as age, sex, pathology, on the questionnaire score by using statistical tests
Measurement of the patients' satisfaction | day 1
  Calculation of the satisfaction rate by using a satisfaction survey
Assess the booklet comprehension | day 1
  number of responses

CONTACTS AND LOCATIONS:
Overall Officials: Christine LEBRUN-FRENAY, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No